CLINICAL TRIAL: NCT04244370
Title: A Prospective, Multi-Center, Single-Arm, Real World Study Assessing the Clinical Use of the Caterpillar™ Arterial Embolization Device for Arterial Embolization in the Peripheral Vasculature (MONARCH)
Brief Title: Caterpillar™ Arterial Embolization Device Post-Market Study
Acronym: MONARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-18-001
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Embolization, Therapeutic
Keywords: Arterial Embolization; Vascular Plug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Caterpillar™ Arterial Embolization Device (Experimental): Placement of the Caterpillar™ Arterial Embolization Device via percutaneous transcatheter embolization (PTE).
  Interventions: Device: Caterpillar™ Arterial Embolization Device

INTERVENTIONS:
Device: Caterpillar™ Arterial Embolization Device — Placement of the Caterpillar™ Arterial Embolization Device for patients requiring arterial embolization in the peripheral vasculature.
  Other Names: Caterpillar™ Micro (027); Caterpillar™ (038 & 056)

SUMMARY:
The primary objective of this study is to evaluate the performance and safety of the Caterpillar™ Arterial Embolization Device when used for arterial embolization in the peripheral vasculature in a real world, on-label application.

DETAILED DESCRIPTION:
The post-market study is a prospective, multi-center, single-arm, real world study of the Caterpillar™ Arterial Embolization Device. Enrollment will continue until up to fifty (50) subjects have been treated with the Caterpillar™ Arterial Embolization Device at up to 20 investigational sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or Legally Authorized Representative (LAR) must voluntarily sign and date the approved Informed Consent Form (ICF) prior to collection of study-specific data or performance of study-specific procedures.
2. Subject must be either male or non-pregnant female ≥18 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
3. Subject must be willing and able to comply with protocol requirements, including all study visits and procedures.
4. Subject must require peripheral vascular occlusion at an arterial target embolization site(s) that can be treated with the Caterpillar™ Arterial Embolization Device according to the Instructions for Use (IFU). Note: Per Investigator discretion, up to five (5) Target Embolization Sites may be treated with up to ten (10) study devices per subject.

   Angiographic Inclusion Criteria
5. The target embolization site(s) must be located in a native arterial vessel(s) with the intended arterial vessel diameter ranges shown in the IFU, as assessed by the Investigator (via visual estimate).
6. The target embolization site(s) must have a landing zone sufficient to accommodate the device implant lengths shown in the IFU.

Exclusion Criteria:

1. The subject's access vessel(s) preclude safe insertion of the delivery catheter.
2. The subject's target embolization site(s) is located within a vein.
3. The subject's target embolization site(s) is located within the head, neck, heart or coronary vessels.
4. The subject's target embolization site(s) is located across highly locomotive joints or muscle beds (e.g. elbow, hip, knee, shoulder, thoracic inlet/outlet).
5. The subject's target embolization site(s) is located in a high-flow vessel where, in the opinion of the Investigator, there may be significant risk of migration and unintended (non-target site) occlusion.
6. The subject has a known allergy or hypersensitivity to contrast media that cannot be adequately pre-medicated.
7. The subject has a known allergy or hypersensitivity to any of the device materials including: cobalt, chromium, nickel, titanium, platinum, iridium, polyurethane or polyethylene.
8. The subject has planned use of anticoagulant (e.g. direct thrombin inhibitors, factor Xa inhibitors, vitamin K antagonists) or antiplatelet therapy before, during and/or after treatment with the study device, which, in the opinion of the Investigator, would clinically interfere with the study endpoints.
9. The subject has a known uncontrolled blood coagulation or bleeding disorder.
10. The subject has an unresolved systemic infection.
11. The subject's required pre-operative laboratory tests and/or physical examination indicate abnormal results, which, in the opinion of the Investigator, would clinically interfere with the study endpoints.
12. The subject has a connective tissue disorders (e.g. Ehlers-Danlos Syndrome), arteritis (e.g. Takayasu's Disease) or another circulatory disorder, which, in the opinion of the Investigator, would clinically interfere with the study endpoints.
13. The subject has another medical condition which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, may confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
14. The subject is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Rilling, MD, FSIR, Principal Investigator — Medical College of Wisconsin
Locations (11):
- United States (11):
  - Dignity Health/St. Joseph's & Medical Center, Phoenix, Arizona
  - Baptist Hospital of Miami, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caterpillar™ Arterial Embolization Device
Started | 50
Completed | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 40
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Successful occlusion of the target embolization site(s) as confirmed by the Investigator via angiographic assessment during the Index Procedure. Technical success will be reported for each target embolization site.
Time Frame: During the Index Procedure
Measure: Count of Units; unit: Target Embolization Sites
Units Other Than Participants: Target Embolization Sites
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites) | 56
Target Embolization Sites | 55

2. Primary Outcome: Freedom From Device-Related SAEs
Description: Freedom from device-related serious adverse events (SAE) through 30-day follow-up.
Time Frame: 30 (-7/+21) Days post Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Participants | 50

3. Secondary Outcome: Time Point of Occlusion
Description: The percentage of target embolization site(s) with occlusion at ≤1, ≤2, ≤3, ≤4, ≤5, ≤10 and >10 minutes post-treatment.
Time Frame: During Index Procedure
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 55
Target Embolization Sites (TESs)
  ≤1 minute | 15
  ≤ 2 minutes | 10
  ≤ 3 minutes | 7
  ≤ 4 minutes | 1
  ≤ 5 minutes | 11
  ≤ 10 minutes | 5
  > 10 minutes | 6

4. Secondary Outcome: Freedom From Recanalization
Description: Freedom from clinically relevant recanalization of the target embolization site(s) through 30-days, 6 and 12-months follow-up as confirmed by the Investigator. Clinically relevant recanalization is defined as recanalization through the study device that requires a re-intervention.
Time Frame: 30 (-7/+21) days, 6 months (±30 days) and 12 months (±30 days) Post Index Procedure
Population: Number of TESs analyzed at 6-Months and 12-Months differs from 30-Day follow-up due to subject discontinuation in the study
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 56
Target Embolization Sites (TESs)
  30-Day Follow-up: number analyzed (Participants) | 49
  30-Day Follow-up | 56
  6-Month Follow-up: number analyzed (Participants) | 26
  6-Month Follow-up: number analyzed (Target Embolization Sites (TESs)) | 43
  6-Month Follow-up | 43
  12-Month Follow-up: number analyzed (Participants) | 20
  12-Month Follow-up: number analyzed (Target Embolization Sites (TESs)) | 31
  12-Month Follow-up | 31

5. Secondary Outcome: Freedom From Acute Migration
Description: Freedom from clinically relevant acute migration of the study device(s) as confirmed by the Investigator via angiographic assessment during the Index Procedure. Clinically relevant migration is defined as migration of the study device from the target embolization site that requires intervention.
Time Frame: During Index Procedure
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 62
Target Embolization Sites (TESs) | 62

6. Secondary Outcome: Freedom From Non-Acute Migration
Description: Freedom from clinically relevant migration of the study device(s) through 30 day, 6 month and 12 month follow-up was reported by the Investigators. Clinically relevant migration is defined as migration of the study device from the target embolization site that requires intervention.
Time Frame: 30 (-7/+21) days, 6 months (±30 days) and 12 months (±30 days) Post Index Procedure
Population: Number of devices analyzed at 6-Months and 12-Months differs from 30-Day follow-up due to subject discontinuation in the study
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Devices) | 62
Devices
  30-Day Follow-up: number analyzed (Participants) | 49
  30-Day Follow-up | 62
  6-Month Follow-up: number analyzed (Participants) | 26
  6-Month Follow-up: number analyzed (Devices) | 47
  6-Month Follow-up | 47
  12-Month Follow-up: number analyzed (Participants) | 20
  12-Month Follow-up: number analyzed (Devices) | 34
  12-Month Follow-up | 34

7. Secondary Outcome: Freedom From Device and/or Procedure-Related Adverse Events
Description: Freedom from device and/or procedure-related adverse events (AE) through 30-days, 6 and 12-months follow-up.
Time Frame: 30 (-7/+21) days, 6 months (±30 days) and 12 months (±30 days) Post Index Procedure
Population: Number of Participants analyzed at 6-Months and 12-Months differs from 30-Day follow-up due to subject discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Participants
  30-Day Follow-up | 42
  6-Month Follow-up: number analyzed (Participants) | 39
  6-Month Follow-up | 31
  12-Month Follow-up: number analyzed (Participants) | 31
  12-Month Follow-up | 23

8. Secondary Outcome: Accuracy of Delivery
Description: Accurate delivery of the study device to the target embolization site as assessed by the Investigator.
Time Frame: During Index Procedure
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 62
Target Embolization Sites (TESs) | 61

9. Secondary Outcome: Ease of Trackability/Deliverability
Description: Ease of study device trackability and deliverability as assessed by the Investigator.
Time Frame: During Index Procedure
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 62
Target Embolization Sites (TESs) | 61

10. Secondary Outcome: Ease of Detachment
Description: Ease of study device detachment as assessed by the Investigator.
Time Frame: During Index Procedure
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 62
Target Embolization Sites (TESs) | 62

11. Secondary Outcome: Acceptability of Visibility Under Fluoroscopy
Description: Acceptability of study device visibility under fluoroscopy as assessed by the Investigator.
Time Frame: During Index Procedure
Measure: Count of Units; unit: Target Embolization Sites (TESs)
Units Other Than Participants: Target Embolization Sites (TESs)
Arm/Group | Caterpillar™ Arterial Embolization Device
Number analyzed (Participants) | 50
Number analyzed (Target Embolization Sites (TESs)) | 63
Target Embolization Sites (TESs) | 59

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Caterpillar™ Arterial Embolization Device
All-Cause Mortality (participants affected / at risk) | 5/50
Serious Adverse Events (participants affected / at risk) | 11/50
Other Adverse Events (participants affected / at risk) | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caterpillar™ Arterial Embolization Device (N=50)
Obstruction Gastric (Gastrointestinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caterpillar™ Arterial Embolization Device (N=50)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator seeking publication shall submit to Sponsor for review a draft of the proposed publication at least 60 days prior to submission of the draft for publication. Sponsor shall have the right to: (i) review and make editorial comments on any such proposed publication; and (ii) make any results from the Study known to its customers and governmental agencies prior to publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04244370/Prot_SAP_000.pdf